CLINICAL TRIAL: NCT05260125
Title: Comparison of the Efficacy of Ultrasound Guided vs Non-guided Suprascapular Nerve Block Treatment in Stroke Patients With Hemiplegic Shoulder Pain.
Brief Title: Comparison of the Efficacy of Ultrasound Guided vs Non-guided Suprascapular Nerve Block Treatment in Stroke Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Serdar Kilinc, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIBU-FTR-SK-01
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Hemiplegia; Stroke
MeSH Terms: conditions — Hemiplegia; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided Suprascapular Nerve Block (Experimental): Ultrasound-guided Suprascapular Nerve Block
  Interventions: Drug: Ultrasound-guided Suprascapular Nerve Block
- Anatomical Landmark-guided Suprascapular Nerve Block (Active Comparator): Anatomical Landmark-guided Suprascapular Nerve Block
  Interventions: Drug: Anatomical Landmark-guided Suprascapular Nerve Block

INTERVENTIONS:
Drug: Ultrasound-guided Suprascapular Nerve Block — For suprascapular nerve block, a solution consisting of 5 ml 2% lidocaine, 1 ml Betamethasone dipropionate + Betamethasone sodium phosphate (6.43 mg/ml + 2.63 mg/ml), 4 ml saline will be used.
  Injections will be applied to patients in a sitting position and arm by the side. A linear probe with a frequency of 7-8 MHz on the SonoScape A8 ultrasound device will be used for suprascapular block under ultrasound guidance. the ultrasound probe was placed in the coronal plane over the suprascapular fossa. Suprascapular fossa was scanned from medial to lateral side to identify suprascapular nerve. After identification, solution of suprascapular nerve block will be injected into the area around the nerve under the scanning with in-plane technique with a 22 gauge 90 mm spinal needle.
  Arms: Ultrasound-guided Suprascapular Nerve Block
Drug: Anatomical Landmark-guided Suprascapular Nerve Block — For suprascapular nerve block, a solution consisting of 5 ml 2% lidocaine, 1 ml Betamethasone dipropionate + Betamethasone sodium phosphate (6.43 mg/ml + 2.63 mg/ml), 4 ml saline will be used.
  Injections will be applied to patients in a sitting position and arm by the side. The suprascapular notch projection will be determined using the anatomical landmark technique defined by Dangoisse et al., and then suprascapular nerve block will be applied with a 22 gauge 90 mm spinal needle to the patients
  Arms: Anatomical Landmark-guided Suprascapular Nerve Block

SUMMARY:
The aim of this study is to compare the effectiveness of ultrasound-guided and non-guided suprascapular nerve block in the treatment of patients with hemiplegic shoulder pain, which is one of the most common post-stroke complications.

DETAILED DESCRIPTION:
Hemiplegic shoulder pain is a general term used to describe shoulder pain that occurs after a stroke. It is one of the complications that significantly affects the rehabilitation of patients.The suprascapular nerve takes up 70% of the sensation of the shoulder joint. For this reason, suprascapular nerve block treatment is applied in the treatment of hemiplegic shoulder pain.In patients with hemiplegic shoulder pain, suprascapular nerve block therapy can be performed under ultrasound guidance or using anatomical landmarks. However, there is no study in the literature comparing the effectiveness of ultrasound-guided and unguided suprascapular nerve block in the treatment of hemiplegic shoulder pain Patients with hemiplegic shoulder pain among the patients who received routine conservative rehabilitation treatment in the physical therapy and rehabilitation clinic with the diagnosis of post-stroke hemiplegia will be included in the study.

Hemiplegic patients aged 25-75 years, with shoulder pain lasting for 3 months and with a Visual Analogue Scale (VAS) value > 3 during passive shoulder joint movement will be included in the study.

Exclusion criteria from the study will be determined as mini mental test score < 24, uncontrolled diabetes, coagulopathy, botulinum toxin administration in the last six months, any injection from the shoulder region in the last six months, and hypersensitivity to injection agents.

It will be organized as a prospective randomized study. It is planned to include 50 patients in the study. Patients will be randomized into two groups in equal numbers, stratified by age and sex.

Patients in group 1 will be applied with ultrasound-guided suprascapular nerve block.

Patients in Group 2 will be applied with suprascapular nerve block using defined anatomical points without ultrasound guidance.

Initially, demographic data, medical history, stroke etiology, duration of stroke, body mass index, hemiplegic side information of the patients will be obtained.

Patients in both groups will be evaluated in terms of shoulder joint range of motion, Visual Analogue Scale, Brunnstrom Stages of Stroke Recovery, Barthel Index, Modified Ashworth Scale, The Beck Depression Inventory before the treatment, at the 1st week, 1st month and 3rd month after the injection.

ELIGIBILITY:
Inclusion Criteria:

* Having hemiplegic shoulder pain for 3 months
* Visual analogue scale score > 3 during passive shoulder joint movement on the hemiplegic side

Exclusion Criteria:

* Mini mental test score <24
* Patients with uncontrolled diabetes, coagulopathy
* Botulinum toxin administration in the past six months,
* Any injection in the shoulder region in the last six months
* Having hypersensitivity to injection agents

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Shoulder Range of Motion | Before suprascapular nerve block
  The range of motion of the hemiplegic shoulder joint will be measured passively with a goniometer in the flexion, abduction, internal rotation and external rotation directions.
Shoulder Range of Motion | 1 week after suprascapular nerve block
  The range of motion of the hemiplegic shoulder joint will be measured passively with a goniometer in the flexion, abduction, internal rotation and external rotation directions.
Shoulder Range of Motion | 4 week after suprascapular nerve block
  The range of motion of the hemiplegic shoulder joint will be measured passively with a goniometer in the flexion, abduction, internal rotation and external rotation directions.
Shoulder Range of Motion | 12 week after suprascapular nerve block
  The range of motion of the hemiplegic shoulder joint will be measured passively with a goniometer in the flexion, abduction, internal rotation and external rotation directions.
Visual Analogue Scale | Before suprascapular nerve block
  Pain was evaluated using a 10 cm long Visual Analogue Scale (VAS) during rest and activity (0 = no pain, 10 = very severe pain).
Visual Analogue Scale | 1 week after suprascapular nerve block
  Pain was evaluated using a 10 cm long Visual Analogue Scale (VAS) during rest and activity (0 = no pain, 10 = very severe pain).
Visual Analogue Scale | 4 week after suprascapular nerve block
  Pain was evaluated using a 10 cm long Visual Analogue Scale (VAS) during rest and activity (0 = no pain, 10 = very severe pain).
Visual Analogue Scale | 12 week after suprascapular nerve block
  Pain was evaluated using a 10 cm long Visual Analogue Scale (VAS) during rest and activity (0 = no pain, 10 = very severe pain).

SECONDARY OUTCOMES:
Barthel Index | Before suprascapular nerve block
  The Barthel index is used to assess activities of daily living. It consists of 10 items: feeding, bathing, grooming, dressing, bowel, bladder, toilet use, transfers, mobility, stairs. Scores range from 0-100. A score of 100 represents complete independence, and a score of 0 represents complete dependence.
Barthel Index | 1 week after suprascapular nerve block
  The Barthel index is used to assess activities of daily living. It consists of 10 items: feeding, bathing, grooming, dressing, bowel, bladder, toilet use, transfers, mobility, stairs. Scores range from 0-100. A score of 100 represents complete independence, and a score of 0 represents complete dependence.
Barthel Index | 4 week after suprascapular nerve block
  The Barthel index is used to assess activities of daily living. It consists of 10 items: feeding, bathing, grooming, dressing, bowel, bladder, toilet use, transfers, mobility, stairs. Scores range from 0-100. A score of 100 represents complete independence, and a score of 0 represents complete dependence.
Barthel Index | 12 week after suprascapular nerve block
  The Barthel index is used to assess activities of daily living. It consists of 10 items: feeding, bathing, grooming, dressing, bowel, bladder, toilet use, transfers, mobility, stairs. Scores range from 0-100. A score of 100 represents complete independence, and a score of 0 represents complete dependence.
Modified Ashworth Scale | Before suprascapular nerve block
  Spasticity in the shoulder will be evaluated according to the Modified Ashworth Scale (MAS). The Modified Ashworth Scale is a 6-point scale. Scores range from 0 to 4, where lower scores represent normal muscle tone and higher scores represent increased degree of spasticity.
Modified Ashworth Scale | 1 week after suprascapular nerve block
  Spasticity in the shoulder will be evaluated according to the Modified Ashworth Scale (MAS). The Modified Ashworth Scale is a 6-point scale. Scores range from 0 to 4, where lower scores represent normal muscle tone and higher scores represent increased degree of spasticity.
Modified Ashworth Scale | 4 week after suprascapular nerve block
  Spasticity in the shoulder will be evaluated according to the Modified Ashworth Scale (MAS). The Modified Ashworth Scale is a 6-point scale. Scores range from 0 to 4, where lower scores represent normal muscle tone and higher scores represent increased degree of spasticity.
Modified Ashworth Scale | 12 week after suprascapular nerve block
  Spasticity in the shoulder will be evaluated according to the Modified Ashworth Scale (MAS). The Modified Ashworth Scale is a 6-point scale. Scores range from 0 to 4, where lower scores represent normal muscle tone and higher scores represent increased degree of spasticity.
Brunnstrom Stages of Stroke Recovery | Before suprascapular nerve block
  Brunnstrom Stages of Stroke Recovery will be used to determine the levels of motor function in the upper extremity and hand.
Brunnstrom Stages of Stroke Recovery | 1 week after suprascapular nerve block
  Brunnstrom Stages of Stroke Recovery will be used to determine the levels of motor function in the upper extremity and hand.
Brunnstrom Stages of Stroke Recovery | 4 week after suprascapular nerve block
  Brunnstrom Stages of Stroke Recovery will be used to determine the levels of motor function in the upper extremity and hand.
Brunnstrom Stages of Stroke Recovery | 12 week after suprascapular nerve block
  Brunnstrom Stages of Stroke Recovery will be used to determine the levels of motor function in the upper extremity and hand.
The Beck Depression Inventory | Before suprascapular nerve block
  The Beck Depression Inventory is a 21-question multiple-choice self-report inventory, used instruments for measuring the severity of depression. Scores from 0 to 9 represent minimal depressive symptoms, scores of 10 to 16 indicate mild depression, scores of 17 to 29 indicate moderate depression, and scores of 30 to 63 indicate severe depression.
The Beck Depression Inventory | 1 week after suprascapular nerve block
  The Beck Depression Inventory is a 21-question multiple-choice self-report inventory, used instruments for measuring the severity of depression. Scores from 0 to 9 represent minimal depressive symptoms, scores of 10 to 16 indicate mild depression, scores of 17 to 29 indicate moderate depression, and scores of 30 to 63 indicate severe depression.
The Beck Depression Inventory | 4 week after suprascapular nerve block
  The Beck Depression Inventory is a 21-question multiple-choice self-report inventory, used instruments for measuring the severity of depression. Scores from 0 to 9 represent minimal depressive symptoms, scores of 10 to 16 indicate mild depression, scores of 17 to 29 indicate moderate depression, and scores of 30 to 63 indicate severe depression.
The Beck Depression Inventory | 12 week after suprascapular nerve block
  The Beck Depression Inventory is a 21-question multiple-choice self-report inventory, used instruments for measuring the severity of depression. Scores from 0 to 9 represent minimal depressive symptoms, scores of 10 to 16 indicate mild depression, scores of 17 to 29 indicate moderate depression, and scores of 30 to 63 indicate severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Serdar kılınç, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)